CLINICAL TRIAL: NCT05581043
Title: Pre-meals of 3-hydroxybutyrate for People With Type 2 Diabetes
Brief Title: Pre-meals of 3-hydroxybutyrate in Type 2 Diabetes
Acronym: PreKetone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Steno Diabetes Center Aarhus, Aarhus University Hospital, Denmark (Unknown); Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: V4_03052022
Record Dates: First submitted 2022-10-04; First posted 2022-10-14 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2022-10

CONDITIONS: Ketosis; Postprandial Hyperglycemia; Glucose Metabolism Disorders (Including Diabetes Mellitus)
MeSH Terms: conditions — Ketosis; Hyperglycemia; Glucose Metabolism Disorders | interventions — 3-Hydroxybutyric Acid

STUDY DESIGN:
Intervention Model Description: We will use a randomized cross-over design to investigate 10 volunteers with T2DM on six different occasions separated with at least one week.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 0 gram 3-OHB 30 minutes before an OGTT (Placebo Comparator): 0 gram 3-OHB 30 minutes before an OGTT
  Interventions: Dietary Supplement: 3-hydroxybutyrate (3-OHB)
- 10 gram 3-OHB 30 minutes before an OGTT (Experimental): 10 gram 3-OHB 30 minutes before an OGTT
  Interventions: Dietary Supplement: 3-hydroxybutyrate (3-OHB)
- 20 gram 3-OHB 30 minutes before an OGTT (Experimental): 20 gram 3-OHB 30 minutes before an OGTT
  Interventions: Dietary Supplement: 3-hydroxybutyrate (3-OHB)
- 40 gram 3-OHB 30 minutes before an OGTT (Experimental): 40 gram 3-OHB 30 minutes before an OGTT
  Interventions: Dietary Supplement: 3-hydroxybutyrate (3-OHB)
- 20 gram 3-OHB 0 minutes before an OGTT (Experimental): 20 gram 3-OHB 0 minutes before an OGTT
  Interventions: Dietary Supplement: 3-hydroxybutyrate (3-OHB)
- 20 gram 3-OHB 60 minutes before an OGTT (Experimental): 20 gram 3-OHB 60 minutes before an OGTT
  Interventions: Dietary Supplement: 3-hydroxybutyrate (3-OHB)

INTERVENTIONS:
Dietary Supplement: 3-hydroxybutyrate (3-OHB) — The aim of this study was therefore to i) investigate the dose/response relationship between 3-OHB servings of 0, 10, 20 and 40 grams 30 minutes before an OGTT and, ii) investigate the role of timing by serving 25 grams of 3-OHB at different timepoints ahead of an OGTT (0, 30 and 60 minutes).

SUMMARY:
Hyperglycemia following meals in patients with type 2 diabetes mellitus (T2DM) is a common problem. Recently, our group found that oral consumption of the ketone metabolite, 3-hydroxybutyrate (3-OHB), effectively stimulates insulin secretion and delays gastric emptying.The aim of this study is to investigate the dose/response relationship between 3-OHB servings of 0, 10, 20 and 40 grams 30 minutes before an OGTT and, ii) investigate the role of timing by serving 20 grams of 3-OHB at different timepoints ahead of an OGTT (0, 30 and 60 minutes)

DETAILED DESCRIPTION:
Hyperglycemia following meals in patients with type 2 diabetes mellitus (T2DM) is a common problem, which can cause discomfort and fatigue but may also lead to diabetic complications. Small servings of macronutrients, especially protein-rich products, before a main meal (= pre-meals) has been shown to significantly lower postprandial glucose excursions in both healthy individuals and patients with T2DM. The reductions are primarily attributed the fact that protein stimulates insulin secretion and delays gastric emptying. The timing and dose of a premeal are essential for the glycemic reductions following a meal 4. Unfortunately, it often requires a rather large amount of protein (> 50 g) to facilitate clinically relevant reductions in postprandial glucose levels and a large protein intake may be unwanted for some patients (i.e., chronic kidney disease). Recently, our group found that oral consumption of the ketone metabolite, 3- hydroxybutyrate (3-OHB), effectively stimulates insulin secretion and delays gastricemptying. We have also shown that 3-OHB inhibits gluconeogenesis 6, which may further contribute to glucose-lowering effects. Two other clinical studies have shown that serving 3- OHB before an oral glucose tolerance test (OGTT) lowered glucose excursions in healthy volunteers and persons with impaired glucose tolerance. There are no current data available about the effect of 3-OHB premeals in T2DM patients, but we have preliminary data from an ongoing trial showing that 30 g of 3-OHB served 40 min before a mixed meal test effectively lowers postprandial glucose levels (around 3 mM) in patients with T2DM. The optimal dose and timing of 3-OHB pre-meals is unknown but important before initiating long-term clinical trials. We hypothesize that pre-melas of 3-OHB will affect postprandialglucose excursions in a time-dependent matter and servings 30 minutes before an OGTT is Deleted: 4 optimal in order to lower postprandial glucose excursions. The aim of this study is therefore to i) investigate the dose/response relationship between 3-OHB servings of 0, 10, 20 and 40 grams 30 minutes before an OGTT and, ii) investigate the role of timing by serving 20 grams of 3-OHB at different timepoints ahead of an OGTT (0, 30 and 60 minutes). The primary endpoint is glucose trajectories following the OGTT. This study will give important insight into the optimal dose and timing for potential future clinical long-term studies in patients with metabolic diseases (i.e., T2DM, obesity)

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Type 2 diabetes diagnosis
* No antiglycemic treatment or monotherapy with metformin

Exclusion Criteria:

* Hba1c > 70
* Severe liver disease (Child-Pugh score >10) or kidney disease (eGFR< 40 ml/min)
* Anemia (Hgb < 6.5 mM)
* History with pancreatitis
* Practicing ketogenic diets (i.e., low-carb diet, fasting regime)
* Inability to understand Danish or English
* Ongoing cancer or other acute/chronic serious diseases (PI will determine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose following the OGTT | Blood samples will be obtained -60, -30, -15, 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes from the OGTT
  Change in blood glucose following the OGTT and compared between the different visits. Incremental change (delta) from baseline to peak. Measured with laboratory kits.

SECONDARY OUTCOMES:
Plasma concentrations of 3-OHB, insulin, C-peptide, glucagon like peptide-1 (GLP-1), cholecystokinin (CCK), acetaminophen, free fatty acids along others. | Blood samples will be obtained -60, -30, -15, 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes from the OGTT
  Incremental change (delta) from baseline to peak in plasma concentrations of 3-OHB, insulin, C-peptide, glucagon like peptide-1 (GLP-1) following the OGGT and compared between the different visits. Measured with laboratory kits.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, Professor, Study Director — Professor
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus, Denmark

REFERENCES:
- [Derived] Bangshaab M, Bengtsen MB, Smedegaard S, Sondergaard E, Moller N, Svart MV, Rittig N. Ketone supplementation dose-dependently lowers postprandial blood glucose, lipid and ghrelin levels in individuals with type 2 diabetes: a randomised crossover study. Diabetologia. 2025 Nov 28. doi: 10.1007/s00125-025-06614-0. Online ahead of print. PMID 41315088